CLINICAL TRIAL: NCT05899660
Title: Impact of Omega-3 Polyunsaturated Fatty Acids on Emotional, Cognitive and Biological Alterations in Alcohol Use Disorder
Brief Title: Impact of Omega 3 in Alcohol Use Disorder
Acronym: W3-AUD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2022/22DEC/502
Record Dates: First submitted 2023-05-15; First posted 2023-06-12 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Alcohol Use Disorder, Severe
Keywords: gut microbiota; Omega 3; metabolomics; Depression; Anxiety; Alcohol craving; Sociability; Cognition; Inflammation; Brain imaging
MeSH Terms: conditions — Alcoholism; Depression; Anxiety Disorders; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Olive oil (Placebo Comparator): Dosage form : capsule Dosage : 1000 mg oleic acid (olive oil) + 3.6 mg D-α-tocopherol (vitamin E) Frequency : 4 capsules per day Duration : 3 months
  Interventions: Dietary Supplement: Placebo Comparator: olive oil
- Omega-3 (Active Comparator): Dosage form : capsule Dosage : 330 mg EPA, 220 mg DHA, 100 mg other n-3 PUFA + 3.6 mg D-α-tocopherol (vitamin E) Frequency : 4 capsules per day Duration : 3 months
  Interventions: Dietary Supplement: Active Comparator: Omega-3

INTERVENTIONS:
Dietary Supplement: Active Comparator: Omega-3 — It is a dietary supplement made of fish oil rich in n-3 PUFA.
  Arms: Omega-3
Dietary Supplement: Placebo Comparator: olive oil — Refined olive oil is the usual placebo used in studies with n-3 PUFA.
  Arms: Olive oil

SUMMARY:
The goal of this clinical trial is to investigate the biological pathways underlying the beneficial effect of omega-3 polyunsaturated fatty acids (n-3 PUFA) on mental health in patients with alcohol use disorder. The main questions this study aims to answer are:

* Can n-3 PUFA improve mood disorders (depression, anxiety), craving for alcohol, cognitive impairments and sociability disorders ?
* Are the beneficial effects of n-3 PUFAs due to a modification of the gut microbiota and/or the inflammatory status?

Participants will :

* take a supplementation of omega-3 or placebo during 3 months
* do a brain MRI
* be interviewed for a dietary anamnesis
* provide blood, stool and saliva samples
* perform psychological tests and neuropsychological tasks

Researchers will compare active comparator (omega-3) with placebo comparator (olive oil) to see if omega-3 can have a beneficial effect on AUD patients.

DETAILED DESCRIPTION:
Alcohol use disorder (AUD) is the most widespread addiction in Belgium and Europe and constitutes a major public health problem with important physical, psychological and economic consequences for the consumer and his family, friends, co-workers.

For several years, the intestinal microbiota has been increasingly studied because it seems to play an indispensable role in the proper functioning of the body. Indeed, it is involved in the regulation of the immune system, metabolic reactions and the nervous system and therefore influences behaviour. The composition of the microbiota is specific to everyone and is influenced by many factors, such as diet, medication and lifestyle.

In the case of AUD, numerous studies have shown that alcohol and its metabolites alter the intestinal microbiota, leading to an increase in inflammation and changes in behaviour.

Nutritional intervention is an encouraging and innovative approach to alcohol addiction therapy. The main aim of this research is to see how a nutritional intervention could improve mood, cognition and social behaviour in AUD patients. The interest will therefore focus on Omega-3. These polyunsaturated fatty acids are found in the diet, mainly in fish oils, and are constituents of the body's cell membranes and perform many physiological functions. They also play an important role in the regulation of inflammation. Studies have shown that Omega-3 supplementation can reduce symptoms of depression and have beneficial effects in autism spectrum disorders, schizophrenia, bipolar disorders and neurodegenerative diseases. They have therefore been widely studied, but their role in social interactions, which is an important factor in many mental illnesses including AUD, has not yet been studied.

The investigators will conduct a randomised, placebo-controlled, double-blind study, testing the impact of Omega-3 supplementation on AUD patients undergoing a detoxification program at the Saint-Luc University Hospital, Brussels, Belgium. 100 patients will be enrolled and the Omega 3/placebo supplementation will last for 3 months. The patients will be tested 3 times: T1 (2nd day of withdrawal), T2 (18th-19th day of withdrawal) and T3 (after 3 months of supplementation). The investigators hope to see a beneficial effect of omega-3 on social, emotional and cognitive deficits as well as brain functioning (fMRI). They will investigate the mechanisms involved, namely, changes in the composition of the gut microbiota, reduction of systemic inflammation, and production of bacterial metabolites with immune or neuroactive properties.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of alcohol use disorder (≥ 4 DSM-5 criteria)
* Patient at the hospital for a 3 week alcohol withdrawal program
* Gender : male and female
* Age : between 18 and 70 years old
* Language : french
* Alcohol consumption less than 48 jours before admission

Exclusion Criteria:

* Presence of another addiction, except for smoking and cannabis use
* Presence of a psychiatric comorbidity (axis 1 DSM-5)
* Current or recent use (< 2 months) of antibiotics, probiotics, fibre supplements
* Current or recent (< 2 months) use of omega-3 supplements
* Current or recent (< 2 months) use of oral anti-coagulants drugs
* Current or recent (< 2 months) double anti-platelet therapy
* Coagulation disorders
* Current or recent (< 1 month) use of non-steroidal anti-inflammatory drugs and glucocorticoids
* Morbid obesity : body mass index > 35 kg.m-2
* Bariatric surgery
* Type I diabetes and type II diabetes not stabilised (i.e. glycated haemoglobin > 7.2 and unstable drug treatments)
* Chronic inflammatory diseases
* Cancer (less than 5 years before admission)
* Presence of cirrhosis (Fibroscan® = F4 and echodoppler performed as part of clinical routine on patient admission)
* Known allergy to fish and seafood
* Any other comorbidity that would be a contraindication to the study in the judgement of the principal investigator

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-06-19 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in depression | On day 2, day 19 and day 90
  Beck Depression Inventory (BDI) (score 0-63) Higher score indicates higher depression level.
Change in anxiety | On day 2, day 19 and day 90
  State-Trait Anxiety Inventory (STAI) (score 20-80) Higher score indicates higher anxiety level.
Change in fatigue | On day 2, day 19 and day 90
  Multidimensional Fatigue Inventory (MFI) (score 20-140) Higher score indicates higher fatigue level.
Change in alcohol craving | On day 2, day 19 and day 90
  Obsessive Compulsive Drinking Scale (OCDS) (score 0-40) Higher score indicates higher craving level.
Change in impulsivity | On day 19 and day 90
  Urgency Premeditation Perseverance Sensation seeking impulsive behavior scale (UPPS) : score of different subscales are calculated : "ugency" (0-48), "lack of premeditation" (0-44), "lack of perseverance" (0-40), "sensation seeking) (0-48).
  Higher score in the different subscales indicates higher impulsivity level.
Change in social anxiety | On day 19 and day 90
  Liebowitz Scale of Social Anxiety (EASL) (score 0-144) Higher score indicates higher social anxiety level.
Change in trauma | On day 19
  Post-traumatic diagnostic scale (PDS-F): calculation of score is complex and described in the related publication
Childhood trauma | On day 19
  Childhood Trauma Questionnaire (CTQ) (28-144) Higher score indicates higher childhood trauma level.
Self-stigma | On day 19
  Self-Stigma in Alcohol Dependence (SSAD) (16-80) Higher score indicates higher self-stigma level.
Change in work memory | On day 2, day 19 and day 90
  Letter Memory Task
Change in inhibition | On day 2, day 19 and day 90
  Stop Signal Task
Change in decision making | On day 19 and day 90
  Fisher Task
Change in facial emotions recognition | On day 19 and day 90
  Facial Emotions Recognition Task (TREF)
Change in visual perspective taking | On day 19 and day 90
  Visual Perspective Taking Task
Sociability | On day 19
  Sociogram
Emotional intelligence | Day 19
  Trait Emotional Intelligence Questionnaire (TEI Que-75) : calculation of score is complex and described in the related publication
Change in social activity | On day 2, day 19 and day 90
  Social Activities Questionnaire (28-196)

SECONDARY OUTCOMES:
Change in markers of microbial translocation | On day 2, day 19 and day 90
  measurement of sCD14, PGRP in blood sample using ELISA kits (pg/mL)
Change in inflammation | On day 2, day 19 and day 90
  Circulating pro- and anti-inflammatory cytokines (TNFa, IL-6, IL-1b, IL-8, IL-10) levels in blood sample Isolation of PBMC to study intracellular inflammatory pathways by RT-qPCR
Change in gut microbiota composition | On day 2, day 19 and day 90
  Analysis of gut microbiota (16S rDNA) by high-throughput sequencing (Illumina)
Intestinal permeability | On day 19
  a duodenal biopsy will be collected and the expression of the tight junctions regulation the intestinal permeability will be analyzed by sectional immunofluorescence and quantitative polymerase chain reaction
Change in omega-3 levels | On day 2, day 19 and day 90
  Omega-3 levels in plasma and red blood cells
Change in diet profile | On day 2, day 19 and day 90
  The dietary anamnesis will consist of a 24-hour recall over 3 days (2 weekdays and 1 weekend day)
Change in brain functioning | On day 2, day 19 and day 90
  Magnetic Resonance Imaging

CONTACTS AND LOCATIONS:
Overall Officials: Philippe de Timary, MD, PhD, Principal Investigator — St Luc academic Hospital and Université Catholique de Louvain; Peter Starkel, MD, PhD, Principal Investigator — St Luc academic Hospital and Université Catholique de Louvain
Locations (1):
- Cliniques universitaires Saint Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hearn, M, Ceschi, G., Brillon, P, Fürst, G., & Van der Linden, M. (2012). A French adaptation of the Post-traumatic Diagnostic scale. Canadian Journal of Behavioural Science, 44, 16-28
- [Background] Petrides KV (2009) Psychometric properties of the trait emotional intelligence questionnaire. In: Stough C, Saklofske DH, Parker JD (eds) Advances in the assessment of emotional intelligence. Springer, New York. 10.1007/978-0-387-88370-0_5